CLINICAL TRIAL: NCT05281458
Title: Postponed or Early Drainage of Peripancreatic Fluid Collections: a Randomized Controlled Multicenter Study
Brief Title: Early Versus Standard Endoscopic Interventions for Peripancreatic Fluid Collections
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Second Affiliated Hospital of Soochow University (Other); Shanghai Jiao Tong University Affiliated Sixth People's Hospital (Other); Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Baiwen Li, Director of Digestive Endoscopy Center, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-114
Record Dates: First submitted 2022-02-19; First posted 2022-03-16 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Acute Pancreatitis; Peripancreatic Fluid Collections; Endoscopic Ultrasound-Guided Drainage; Pancreatic Fluid Collections
Keywords: Acute Pancreatitis; Peripancreatic Fluid Collections; Endoscopic Ultrasound; Endoscopic Drainage
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early endoscopic interventions for AP (Experimental): Participants in the intervention group will undergo EUS guided drainage earlier (≤1 weeks) in the disease course.
  Interventions: Procedure: Early drainage of peripancreatic fluid collections
- Standard endoscopic interventions for AP (No Intervention): Participants in the control group will have postponed drainage, preferably until AP progress to the walled-off necrosis stage.

INTERVENTIONS:
Procedure: Early drainage of peripancreatic fluid collections — Participants will undergo EUS guided drainage earlier (≤1 weeks) in the disease course.
  Arms: Early endoscopic interventions for AP

SUMMARY:
Acute pancreatitis is a complex gastrointestinal disease with a variable course that is often difficult to predict early in its development. The majority of cases are mild, self-limited, and follow an uncomplicated course. However, 10-20% of cases can be associated with pancreatic or peripancreatic fluid collections, or both. Infected necrosis complicates 10% of all acute pancreatitis episodes and is associated with a mortality of 15-20%. Current guidelines for necrotizing pancreatitis recommend to postpone drainage until 4 or more weeks after initial presentation to allow collections to "walled-off". However, evidence of infection with clinical deterioration despite maximum support may mandate earlier intervention. It is unclear whether such delay is needed for drainage or whether earlier endoscopic intervention could actually be beneficial in the current approach. The aims of this randomized, controlled, multicenter study is to evaluate whether early endoscopic drainage in patients with peripancreatic fluid collection is superior to postponed intervention in the current practice.

DETAILED DESCRIPTION:
EUS guided drainage is now the preferred route for peripancreatic fluid collections (PFC). It belongs to transmural drainage and is accomplished by creating a fistula and placing a stent between the gastric or duodenal lumen and the PFC. The size of the PFC and percentage of solid debris were noted prior to puncture, and the optimal site of transluminal puncture was identified using EUS. Participants will be randomly allocated to either the intervention or the control group. Participants in the intervention group will undergo EUS guided drainage earlier (≤1 weeks) in the disease course. The follow-up duration is 6 months from randomization. All patients undergo imaging (contrast enhanced computed tomography) at 3- and 6-months post randomization.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with PFC;
* All patients with PFC will be screened for eligibility including a protocolized approach;
* Patients admitted within 72 hours of onset

Exclusion Criteria:

* More than 30 days after onset of acute pancreatitis
* Pregnant women
* Documented chronic pancreatitis
* Inability to gave informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-09-15 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Changes in the Bedside Index of Severe Acute Pancreatitis (BISAP) | 1-4 week
  Comparison of BISAP changes between the two groups after different treatments. Also compare the number of participants with BISAP ≥3. BISAP was designed as a predictor of mortality based on 5 variables: blood urea nitrogen (BUN) level greater than 25 mg/dL, impaired mental status, systemic inflammatory response syndrome (SIRS), age older than 60 years, or radiographic evidence of pleural effusion within the first 24 hours of admission. A BISAP score of 3 or greater was associated with developing organ failure, and a higher scores mean a worse outcome.
Number of Participants with New-onset multi-organ failure after intervention | 1-4 week

SECONDARY OUTCOMES:
Rates of mortality | 6 months
Length of hospital stay | 3 months
Length of ICU stays | up to 3 months
Related complications | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai General Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hines OJ, Pandol SJ. Management of severe acute pancreatitis. BMJ. 2019 Dec 2;367:l6227. doi: 10.1136/bmj.l6227. PMID 31791953
- [Background] Zerem E, Imamovic G, Susic A, Haracic B. Step-up approach to infected necrotising pancreatitis: a 20-year experience of percutaneous drainage in a single centre. Dig Liver Dis. 2011 Jun;43(6):478-83. doi: 10.1016/j.dld.2011.02.020. Epub 2011 Apr 8. PMID 21478061
- [Background] Mallick B, Dhaka N, Gupta P, Gulati A, Malik S, Sinha SK, Yadav TD, Gupta V, Kochhar R. An audit of percutaneous drainage for acute necrotic collections and walled off necrosis in patients with acute pancreatitis. Pancreatology. 2018 Oct;18(7):727-733. doi: 10.1016/j.pan.2018.08.010. Epub 2018 Aug 21. PMID 30146334
- [Background] Hongyin L, Zhu H, Tao W, Ning L, Weihui L, Jianfeng C, Hongtao Y, Lijun T. Abdominal paracentesis drainage improves tolerance of enteral nutrition in acute pancreatitis: a randomized controlled trial. Scand J Gastroenterol. 2017 Apr;52(4):389-395. doi: 10.1080/00365521.2016.1276617. Epub 2017 Jan 4. PMID 28050922
- [Background] Baron TH, DiMaio CJ, Wang AY, Morgan KA. American Gastroenterological Association Clinical Practice Update: Management of Pancreatic Necrosis. Gastroenterology. 2020 Jan;158(1):67-75.e1. doi: 10.1053/j.gastro.2019.07.064. Epub 2019 Aug 31. PMID 31479658
- [Background] Trikudanathan G, Tawfik P, Amateau SK, Munigala S, Arain M, Attam R, Beilman G, Flanagan S, Freeman ML, Mallery S. Early (<4 Weeks) Versus Standard (>/= 4 Weeks) Endoscopically Centered Step-Up Interventions for Necrotizing Pancreatitis. Am J Gastroenterol. 2018 Oct;113(10):1550-1558. doi: 10.1038/s41395-018-0232-3. Epub 2018 Oct 2. PMID 30279466
- [Background] Liu RH, Wen Y, Sun HY, Liu CY, Zhang YF, Yang Y, Huang QL, Tang JJ, Huang CC, Tang LJ. Abdominal paracentesis drainage ameliorates severe acute pancreatitis in rats by regulating the polarization of peritoneal macrophages. World J Gastroenterol. 2018 Dec 7;24(45):5131-5143. doi: 10.3748/wjg.v24.i45.5131. PMID 30568390
- [Background] Rana SS, Verma S, Kang M, Gorsi U, Sharma R, Gupta R. Comparison of endoscopic versus percutaneous drainage of symptomatic pancreatic necrosis in the early (< 4 weeks) phase of illness. Endosc Ultrasound. 2020 Nov-Dec;9(6):402-409. doi: 10.4103/eus.eus_65_20. PMID 33318376
- [Background] Banks PA, Bollen TL, Dervenis C, Gooszen HG, Johnson CD, Sarr MG, Tsiotos GG, Vege SS; Acute Pancreatitis Classification Working Group. Classification of acute pancreatitis--2012: revision of the Atlanta classification and definitions by international consensus. Gut. 2013 Jan;62(1):102-11. doi: 10.1136/gutjnl-2012-302779. Epub 2012 Oct 25. PMID 23100216
- [Background] Mederos MA, Reber HA, Girgis MD. Acute Pancreatitis: A Review. JAMA. 2021 Jan 26;325(4):382-390. doi: 10.1001/jama.2020.20317. PMID 33496779